CLINICAL TRIAL: NCT03948035
Title: Elotuzumab in Combination With Carfilzomib, Lenalidomide and Dexamethasone (E-KRd) Versus KRd Prior to and Following Auto-SCT in Newly Diagnosed Multipe Myeloma and Subsequent Maintenance With Elotuzumab and Lenalidomide Versus Single-Agent Lenalidomide- A Phase III Study by DSMM
Brief Title: Elotuzumab in Combination With Carfilzomib, Lenalidomide and Dexamethasone (E-KRd) Versus KRd in MM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: ClinAssess GmbH (Industry); Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSMM XVII; 2017-001616-11 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2019-05-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: multiple myeloma; autologous stem cell transplant; Elotuzumab; Carfilzomib; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; carfilzomib; Lenalidomide; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-KRd/ Arm A (Experimental): Induction/ Consolidation: Elotuzumab, Carfilzomib, Lenalidomide, Dexamethasone (E-KRd), autologous stem cell transplant, Maintenance: Elotuzumab, Lenalidomide
  Interventions: Drug: Elotuzumab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone; Other: autologous stem cell transplant
- KRd/ Arm B (Active Comparator): Induction/ Consolidation: Carfilzomib, Lenalidomide, Dexamethasone (KRd), autologous stem cell transplant, Maintenance: Lenalidomide
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone; Other: autologous stem cell transplant

INTERVENTIONS:
Drug: Elotuzumab — i.v. infusion. Induction 6 cycles: 10mg/kg BW D1,8,15,22 of cycle 1 and 2, D1,15 of cycles 3-6. Consolidation 4 cycles: 10mg/kg BW D1,15 of cycle 1-4. Maintenance 28-day cycles: 20mg/kg BW D1 of each 28-day cycle.
  Other Names: Empliciti®
  Arms: E-KRd/ Arm A
Drug: Carfilzomib — i.v. infusion. Induction 6 cycles: 20 mg/m² on D1 and 2 of cycle 1, 36 mg/m² on D8, 9, 15, 16 of cycle 1, 36 mg/m² on D1,2,8,9,15,16 of cycle 2-6; Consolidation 4 cycles: 36 mg/m² on days 1, 2, 8, 9, 15, 16 of cycles 1-4.
  Other Names: Kyprolis®
Drug: Lenalidomide — hard capsule for oral use. Induction 6 cycles: 25mg D1-21 of cycle 1-6. Consolidation 4 cycles: 15mg D1-21 of cycle 1, 25mg D1-21 ov cycle 2-4. Maintenance 28-day cycles: 10mg D1-28 of cycle 1,2,3, 15mg D1-28 of cycle 4 and all subsequent cycles.
  Other Names: Revlimid®
Drug: Dexamethasone — orally and i.v. IN ARM A:Induction 6 cycles: 28mg p.o. and 8mg i.v. D1,8,15,22 of cycles 1-2 and D1,15 of cycles 3-6, 40mg p.o. D8,22 of cycle 3-6. Consolidation 4 cycles: 28mg p.o. and 8mg i.v. D1,15 of cycle 1-4 and 20mg p.o. D8,22 of cycle 1-4. IN ARM B: Induction 6 cycles: 40mg p.o. D1,8,15,22 of cycles 1-6. Consolidation 4 cycles: 20mg p.o. D1,8,15, 22 of cycle 1-4 .
  Other Names: Fortecortin®
Other: autologous stem cell transplant — autologous stem cell transplant

SUMMARY:
Of the next-generation compounds, the monoclonal antibodies (moAbs) have recently attracted a lot of interest in MM. The anti-SLAMF7 directed moAb elotuzumab has completed phase III trials in MM patients. One phase III trial in MM patients with one to three prior lines of therapy compared elotuzumab-Rd with standard Rd. The triple combination was shown to significantly prolong PFS in this patient cohort with a greater proportion of patients in at least very good partial response (VGPR) when compared to subjects on Rd. Notably, the rate of infusion-related reactions with this specific moAb was very low, with an overall rate of 10% in premedicated patients and only 1% of Grade 3 severity. Grades 4/5 infusion-related reactions were absent and only 1% of patients on elotuzumab discontinued for infusion-related reactions. Of particular interest is the observation in this trial, that response and PFS were independent of cytogenetic high-risk features, i.e., deletion of chromosome 17p and translocation t(4;14). This effect distinguishes elotuzumab from most, if not all, other drug-based approaches.

The investigators assume that incorporating the moAb into the KRd triple induction regimen should result in an even higher rate of deep (negative for MRD in conjunction with at least very good partial response [VGPR] as defined by the International Myeloma Working Group [IMWG]) with these responses occurring independently of cytogenetic risk. Due to potential interference of elotuzumab with serum immune fixation, the investigators chose VGPR rather than complete response (CR) to exclude false-positive immunofixation results. Furthermore the investigators hypothesize that combining elotuzumab with lenalidomide should prolong PFS further.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a cancer originating from the antibody-secreting plasma cell and characterized by abnormal accumulation of clonal plasma cells in bone marrow. In Europe, 3.8 new cases of MM and 2.2 deaths per 100,000 individuals (age-standardized rate) due to MM were estimated in 2012.

Treatment options for myeloma patients have markedly improved during the last decades.

For frontline treatment, high-dose myeloablative chemotherapy followed by reinfusion of autologous peripheral blood stem cells has been a standard of care since 1996. Introduction of the proteasome inhibitor bortezomib and the immunomodulatory drugs thalidomide and lenalidomide led to improvement in remission rates and survival in newly diagnosed patients. However, high-dose chemotherapy remains essential for achievement of long-lasting remissions even in the era of novel agents.

While high-dose melphalan chemotherapy (HDT) plus autologous stem cell transplant (ASCT) remains a standard in eligible, medically fit subjects, defining an optimal pre- and post HDT approach is subject to rapidly evolving novel-compound based options. In 2010, a group from the U.S. presented results on the combination of lenalidomide, bortezomib, and dexamethasone (VRd) in newly diagnosed patients with an overall response rate of 98%, however without systematic consolidation by HDT. The next-generation proteasome inhibitor carfilzomib is more active and very well tolerated in terms of peripheral neuropathy and gastrointestinal adverse effects. A randomized phase III trial in pretreated myeloma patients found the triple regimen of carfilzomib and lenalidomide/dexamethasone (Rd) to be superior to standard-Rd in terms of depth of response; progression-free survival (PFS) and, most importantly, overall survival (OS). At the 2015 annual meetings of the American Society of Clinical Oncology as well as the European Society of Hematology, this regimen (KRd) was found to be exceptionally effective in a phase 2 trial when given in newly diagnosed patients in a prolonged fashion: patients received four KRd induction cycles prior to HDT. The latter was followed by an additional 4 consolidation and 8 maintenance cycles with KRd, followed by lenalidomide maintenance thereafter. The most appealing effect was the high rate of deep remissions: stringent complete response (sCR) rate increased from 22% following 4 x KRd and HDT to more than 80% following all 18 cycles. Notably, the vast majority of patients in sCR also were negative for minimal residual disease (MRD) as assessed by 10-color flow cytometry. MRD negativity probably has a major impact on long-term disease control as was recently shown in a French prospective trial investigating in the combination of VRd prior and post HDT followed by lenalidomide maintenance.

Of the next-generation compounds, the monoclonal antibodies (moAbs) have recently attracted a lot of interest in MM. The anti-SLAMF7 directed moAb elotuzumab has completed phase III trials in MM patients. One phase III trial in MM patients with one to three prior lines of therapy compared elotuzumab-Rd with standard Rd. The triple combination was shown to significantly prolong PFS in this patient cohort with a greater proportion of patients in at least very good partial response (VGPR) when compared to subjects on Rd. Notably, the rate of infusion-related reactions with this specific moAb was very low, with an overall rate of 10% in premedicated patients and only 1% of Grade 3 severity. Grades 4/5 infusion-related reactions were absent and only 1% of patients on elotuzumab discontinued for infusion-related reactions. Of particular interest is the observation in this trial, that response and PFS were independent of cytogenetic high-risk features, i.e., deletion of chromosome 17p and translocation t(4;14). This effect distinguishes elotuzumab from most, if not all, other drug-based approaches.

The investigators assume that incorporating the moAb into the KRd triple induction regimen should result in an even higher rate of deep (negative for MRD in conjunction with at least very good partial response [VGPR] as defined by the International Myeloma Working Group [IMWG]) with these responses occurring independently of cytogenetic risk. Due to potential interference of elotuzumab with serum immune fixation,the investigators chose VGPR rather than complete response (CR) to exclude false-positive immunofixation results. Furthermore the investigators hypothesize that combining elotuzumab with lenalidomide should prolong PFS further.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for autologous stem cell transplantation (ASCT)
* Patient must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma (only dexamethasone at a cumulative dose of 320 mg; plasmapheresis/dialysis without concomitant chemotherapy,local irradiation of bone lesions; and surgical intervention permitted as pretreatment)
* Newly diagnosed multiple myeloma according to the IMWG updated criteria42: Clonal bone marrow plasma cells ≥ 10% or biopsy proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events:
* Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

  * Hypercalcaemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * Renal insufficiency: creatinine clearance < 40 mL per min or serum creatinine > 177 μmol/L (> 2 mg/dL)
  * Anaemia: haemoglobin value of > 2 g/dL below the lower limit of normal, or a haemoglobin value < 10 g/dL
  * Bone lesions: one or more osteolytic lesions on skeletal radiography,computed tomography (CT), or PET-CT
* Any one or more of the following markers of malignancy:

  * Clonal bone marrow plasma cell percentage ≥ 60%
  * Involved: uninvolved serum free light chain ratio ≥ 100, provided the absolute level of the involved light chain is at least 100 mg/L
  * One or more focal lesions of at least 5mm or greater in size on MRI studies
* Measurable disease parameters as follows:
* Serum monoclonal paraprotein (M-component) level ≥ 1 g/dL and/or urine M-protein level ≥ 200 mg/24 hours or
* In case of IgA myeloma: Serum monoclonal paraprotein level ≥ 0.5 g/dL and/or urine M-protein level ≥ 200 mg/24 hours or
* For patients with no detectable M-component: Serum FLC Assay: Involved FLC level ≥ 10 mg/dL (≥ 100 mg/L) provided serum FLC ratio is abnormal
* ECOG Performance Status ≤ 2
* Laboratory test results within these ranges:
* White blood cell count ≥ 2 x 109/L
* Absolute neutrophil (ANC) count ≥ 1.0 x 109/L
* Platelet count ≥ 75 x 109/L
* Haemoglobin > 8 g/dL
* Calculated creatinine clearance (according to MDRD) ≥ 30 mL/minute
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST and ALT ≤ 2.5 x ULN
* Corrected serum calcium level < 3.5 mmol/L (< 14 mg/dL)
* Patient's legal capacity to consent to study participation
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study has been obtained.
* All females

  * must acknowledge to have understood the hazards lenalidomide can cause to an unborn fetus and the necessary precautions associated with the use of lenalidomide.
  * must use adequate contraception and agree to use two reliable forms of contraception simultaneously or to practice complete abstinence
  * must agree to have medically supervised pregnancy tests on a regular basis
  * must agree to abstain from breastfeeding while taking lenalidomide, carfilzomib and elotuzumab and for at least 28 days after the last dose of lenalidomide, carfilzomib, and elotuzumab.
* Male subjects must

  * practice complete abstinence or use a condom during sexual contact with a pregnant female or a female with child bearing potential while taking lenalidomide, carfilzomib, and elotuzumab.
  * not donate semen or sperm
* All subjects must

  * agree to abstain from donating blood while taking lenalidomide, during dose interruptions and for at least 28 days after the last dose of lenalidomide.
  * agree never to give lenalidomide to another person.
  * agree to return all unused lenalidomide capsules to the investigator (with exception of prescribed lenalidomide capsules)
  * be aware that no more than a 28-day lenalidomide supply may be dispensed with each cycle of lenalidomide during induction and consolidation therapy and be prescribed during maintenance therapy.

Exclusion Criteria:

* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy,
* monoclonal protein, and skin changes)
* Waldenström's macroglobulinemia or IgM myeloma
* Plasma cell leukemia (> 2.0 x 109/L circulating plasma cells by standard differential blood count)
* Pregnant, breast-feeding females, FCBPs and males who are unwilling to comply with the lenalidomide Pregnancy Prevention Risk Management Plan.
* Patients with high cardiovascular risk, including but not limited to history of myocardial infarction or coronary stenting in the past 6 months; NYHA Class III or IV heart failure, uncontrolled angina, uncontrolled hypertension, severe uncontrolled arrhythmias
* Prior cerebral vascular accident (CVA) with persistent neurological deficit
* Active infection
* Known HIV-seropositivity, active or chronic hepatitis A, B, C or D-infection (including patients who are tested anti-HBC positive and/or HBsAg positive).
* Any other severe concomitant disease or disorder, including the presence of laboratory abnormalities, which places the subject at unacceptable risk or which could influence patient's ability to participate in the study and his/her safety during the study or interfere with interpretation of study results.
* Greater or equal to Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment
* Major surgery within 4 weeks prior to randomization
* Any systemic anti-myeloma therapy within 4 weeks of randomization except a max. cumulative dose of 320 mg auf dexamethasone.
* Any prior or concurrent malignancy other than multiple myeloma.
* Exceptions include patients who have been disease-free for at least five years before study entry or patients with adequately treated and completely resected basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer.
* Known hypersensitivity to carfilzomib, lenalidomide, and elotuzumab or to any of the excipients of carfilzomib, lenalidomide, and elotuzumab or to any other component of any study drug formulation
* Participation in any other clinical trial or treatment with any experimental drug or other experimental therapy within 28 days before enrolment to the study or during study participation until the end of treatment visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Induction phase | At the end of Cycle 6 (168 days for all cycles plus up to 36 days)
  MRD negativity rate (%) as assessed by flow-cytometry in patients with VGPR or better response according to IMWG criteria following six cycles of induction treatment.
Maintenance phase | 3 years from randomisation
  Determination of progression-free survival (PFS) following randomisation

SECONDARY OUTCOMES:
Measurement of long-term efficacy (1) | 10 years
  Overall response rate (%) to treatment
Measurement of long-term efficacy (2) | 10 years
  Overall survival (months)
Measurement of long-term efficacy (3) | 10 years
  Quality of Life (Units on Scale; Unit range from 0 to 100; Units calculated via linear transformation of raw score (RS) values from scale with single-item measure from 1 to 7 on EORTC QLQ-C30 questionnaire equivalent; Formular for transformation: Unit = {(RS-1)/6}x100)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Einsele, MD, Principal Investigator — Wuezburg University Hospital
Locations (56):
- Austria (10):
  - Univ. Klinikum Krems, Krems, Lower Austria
  - Universitätklinikum St. Pölten, Sankt Pölten, Lower Austria
  - LKH-Universitätsklinikum Graz, Graz, Styria
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Kepler Universitätsklinikum, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - LKH Rankweil-Feldkirch, Rankweil, Vorarlberg
  - Landeskrankenhaus Salzburg, Salzburg
  - AKH Meduni Wien, Vienna
  - Klinik Ottakring, Vienna
- Germany (46):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Kliniken Ostalb, Mutlangen, Baden-Wurttemberg
  - Studienzentrum Onkologie Ravensburg, Ravensburg, Baden-Wurttemberg
  - Diakonieklinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Robert-Bosch Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Onkologie Schwarzwald-Alb, Villingen-Schwenningen, Baden-Wurttemberg
  - Gesundgheitszentrum St. Marien, Amberg, Bavaria
  - Klinikum Augsburg, Augsburg, Bavaria
  - Sozialstiftung Bamberg, Bamberg, Bavaria
  - Klinikum Bayreuth, Bayreuth, Bavaria
  - Klinikum Kempten-Oberallgäu, Kempten (Allgäu), Bavaria
  - Rotkreuzklinikum München, Munich, Bavaria
  - Ludwig-Maximilians-Universität München, Munich, Bavaria
  - Klinikum rechts der Isar der TU München, Munich, Bavaria
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Uniklinikum Regensburg, Regensburg, Bavaria
  - Klinikum Traunstein, Traunstein, Bavaria
  - Universitätsklinikum Würzburg, Medizinische Klinik II, Würzburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main, Hesse
  - Universitätsklinikum Göttingen, Göttingen, Lower Saxony
  - Med. Hochschule Hannover, Hanover, Lower Saxony
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Universitätmedizin Greifswald, Greifswald, Mecklenburg-Pomerania
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Pomerania
  - Helios Kliniken, Schwerin, Mecklenburg-Pomerania
  - Evangelisches Klinikum Bethel, Bielefeld, North Rhine-Westphalia
  - St. Johannes Hospital, Dortmund, North Rhine-Westphalia
  - St. Barbara-Klinik Hamm, Hamm, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - St. Marien-Krankenhaus, Siegen, North Rhine-Westphalia
  - Gemeinschaftsklinikum Mittelrhein, Koblenz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Malteser Krankenhaus, Flensburg, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Zentralklinik Bad Berka, Bad Berka, Thuringia
  - Klinikum der Friedrich-Schiller-Universität Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Helios Kliniken, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Asklepios Klinik Altona, Hamburg

REFERENCES:
- [Derived] Rassner M, Baur R, Wasch R, Schiffer M, Schneider J, Mackensen A, Engelhardt M. Two cases of carfilzomib-induced thrombotic microangiopathy successfully treated with Eculizumab in multiple myeloma. BMC Nephrol. 2021 Jan 18;22(1):32. doi: 10.1186/s12882-020-02226-5. PMID 33461512